CLINICAL TRIAL: NCT04054258
Title: Effectiveness of the Nurse-led Support Programme Using a Mobile Application Versus Telephone Advice on Patients at Risk of Coronary Heart Disease - a Pilot Randomized Controlled Trial
Brief Title: Program Using a Mobile Application Versus Telephone Advice on Patients at Risk of Coronary Heart Disease : a Pilot RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Eliza Wong, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16172411
Record Dates: First submitted 2019-08-05; First posted 2019-08-13 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Coronary Heart Disease
Keywords: coronary heart disease; e-health; self-efficacy
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Intervention Model Description: A prospective multi-center, parallel, randomized controlled trial with two arms: app support (ASP) group v.s. a telephone support (TS) group. Two-Armed study design may yield reliable evidence about the interventional use of app support v.s. telephone support, and will allow us to directly investigate the cause and effects. This design is guided by the CONSORT checklist.
Who Masked: Participant
Masking Description: Randomization will be 1:1 to each treatment arm and will be stratified by the center. Block randomization with varying block sizes will be used to recruit equal numbers to each arm. A computer-generated randomizer will be used to generate the random allocation list. A statistician (DL) from the research team who is not involved in recruiting patients or collecting data will perform the randomization. Each eligible subject will be assigned a number generated by the computer. Subjects will be randomly allocated to different groups according to their number. In this study, the statisticians, outcome assessors, and research assistants assigned to perform data inputting will be blinded to the allocation sequence. Given the type of intervention, however, the intervention will be unmarked to the participants and the research nurse performing the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App support programme group (Experimental): In addition to the usual care, the participant and one family member will receive a CHD app and a briefing from a trained research nurse (A). The reason to invite an additional family member to install the app is to ensure that he/she can be informed automatically when the patient presses an icon during a chest pain attack. The patient may be too stressed during an angina attack and may not be able to follow the 'Things to Do List' quickly. In addition, automatic reminders of the individual's medication times and follow-up times will be pre-set in the app for individual use.
  Interventions: Device: App support Programme (ASP) group
- Telephone support group (Active Comparator): In addition to the above usual care, bi-weekly 20-minute telephone follow-ups will be provided by a trained research nurse (B) for up to 3 months. Patients can ask about related health problems if any. The nurse will address their problem by providing advice or referring them to the ED follow-up clinic. The team has set up a telephone advice guide to support the research nurse in giving phone advice.
  Interventions: Device: App support Programme (ASP) group

INTERVENTIONS:
Device: App support Programme (ASP) group — All subjects will continue their usual care with prescribed medical treatments, ED nursing advice, and follow-ups as indicated. In addition to the above usual care, bi-weekly 20 minutes telephone follow ups will be provided by a trained research nurse (B) up to 3 months. Patients can ask related health problems if any. The nurse will address their problem by providing advices or refer them to the ED follow up clinic if the problems cannot be solved by the nurse.
  Other Names: Telephone support group

SUMMARY:
Topic: Effectiveness of the nurse-led support programme using a mobile application versus telephone advice on patients at risk of coronary heart disease - a randomized controlled trial

Aims: The study aims to compare the effects of a nurse-led support programme using a mobile application versus telephone advice on patients at risk of coronary heart disease who have been discharged from the emergency department (ED).

Methods: A multi-centre, single-blinded, randomized controlled trial will be conducted. 80 patients diagnosed as being at risk of CHD, able to use a smart phone, and who have been discharged from the ED will be randomized into the App Support Programme (ASP) group or the Telephone Support (TS) group. All participants will receive standard medical and nursing care on discharge. The ASP group will receive an app whereas the TS group will receive telephone support provided by the nurse for 20 minutes bi-weekly.

The self-developed mobile app will support clients in managing their health problems and lifestyle. It is comprised of: (1) a knowledge health platform, (2) a membership area for individual health measures and exercise records, (3) a Chest Pain - Things to Do List, and (4) an individual reminder and measure feedback system.

Health outcomes will be collected at baseline (T0), 1 month (T1), 3 months (T2). The primary outcome is Self-efficacy and self-management behavior. Secondary outcomes are: (i) ED and hospitalization frequency; (ii) Physiological health profile and cardiovascular functional endurance; (3) total amount of exercise; (4) perceived stress level; (5) health literacy; and (6) quality of life.

Data analysis: A Generalized Estimating Equations model will be used to assess differential changes in all outcome variables.

DETAILED DESCRIPTION:
Aims and Hypotheses to be Tested:

This study compares the effects of a nurse-led support programme - an app support programme (ASP) - with telephone support (TS) for patients discharged from the ED who are at risk of developing CHD. We hypothesize that:

Within 3 months, when compared with the TS group clients, clients who participate in the ASP will have:

Primary outcome: Better self-efficacy and self-management behaviour

Secondary outcomes:

* Less ED attendance and hospitalization frequency;
* A better physiological health profile (e.g., blood pressure, body mass index, blood cholesterol level, blood triglyceride level, and blood glucose level) and better cardiovascular functional endurance;
* An increase in the total amount of exercise;
* A lower perceived stress level; and
* Better health literacy regarding cardiac care.

Plan of Investigation:

(i)Methods: A prospective multi-center, parallel, randomized controlled trial with two arms - an app support programme (ASP) group vs a telephone support (TS) group - will be adopted. 1. Settings: Data will be collected from an EDs at a regional Hong Kong hospital, namely Tuen Mun Hospital and the community centres. The demographic profile of the residents and the setting and care protocol will be similar, to minimize the cluster effect. Each ED includes a short stay unit and an emergency medical unit (EMW) with about 26 beds. Patients with cardiac disorders account for approximately 25% of all EMW admissions (n=1900 per year) and generally have hypertension or hyperlipidemia and angina 4.

2. Recruitment of subjects: The admission records of all eligible clients with a medical diagnosis of at-risk CHD in the study ED will be screened. Identified patients will be approached by the research assistant (RA1) for further screening and those deemed to be eligible will be invited to join the study. Appendix 2 presents the CONSORT flow diagram of the study.

About 80 potential patients will be approached. Eligible patients who consent to participate in the study and then who submit to the collection of their baseline data will be randomly allocated to either the ASP group or the TS group according to the pre-set randomization sequence. Participants will attend an appointment with a research nurse (A) who has experience in cardiac nursing and specific training in the intervention. Follow-ups will be conducted at 1 month, and 3 months by another RA (2), who will be blinded to the intervention allocation.

Regarding patient recruitment, we estimate that 75% of eligible CHD patients (n=5-7 per week) will agree to join the study at an ED and that at least 8-10 patients will be recruited from both EDs per week. These estimations are based on local departmental statistics and on a previous study that we conducted in a regional ED. 4 We further estimate that 10 weeks will be required to recruit all of the patients required for the study (60 patients). Due to the Covid- 19 situation that subject recruitment is not allowed, we also extend the subject recruitment to community centres..Subject inclusion criteria are the same. Ethical approval has been obtained from the university and the study venues.

3. Follow-up data collection: During the 1-, and 3-month follow-ups, the trained RA (2) and student research assistants (who are master's nursing students), who will be blinded to group allocation, will collect data and perform physical assessments of the participants at the university's research laboratory office. This office has sufficient space and equipment to perform health assessments and laboratory tests. "Item e" shows the facilities in detail. All participants will be asked to complete the questionnaires, place them in an envelope, and hand the envelope to the research assistants.

To ensure the quality of patient recruitment, intervention, and data collection processes, the research team will ensure that the RAs and research nurses are capable of carrying out the proper procedures. All of the research nurses are qualified and experienced in cardiac nursing. They will be provided with specific training workshops by the PI and Co-Is prior to the commencement of the study. One research nurse (A) who is skilled in cardiac nursing and counseling will deliver all of the educational interventions to ensure consistency. Audit procedures will be conducted to ensure the quality and uniformity of the educational intervention. Another research nurse (B) will provide the telephone advice intervention to the TSG. The team will visit the EDs at least once per week during the initial recruitment period. Weekly meetings with research nurses and research assistants will be held to ensure good quality in data collection and to solve any logistical problems.

Data processing and analysis To minimize subject contamination, the different groups will be assigned different follow-up dates. The research assistants who are responsible for collecting data will be blinded to the group allocations. They will receive a briefing and training session on collecting data, taking blood using the finger-stick method, and using the auto blood analyzers. All questionnaires will be distributed to the individual participants, who will be asked to place their own completed questionnaire in a locked box.

Data will be analyzed using SPSS. The intention-to-treat principle will be applied. The baseline characteristics of the groups will be compared using a Chi-square or Fisher's exact test for categorical variables, and a t-test or Mann-Whitney test for continuous variables, to examine the comparability of the groups by randomization. Confounding variables will be accounted for in subsequent analyses. The effectiveness of an e-health programme using the app vs telephone support will be evaluated by comparing the study outcomes using Generalized Estimating Equations (GEE) models. For the primary outcomes of self-efficacy and self-management behavior, two GEE models with an identity link function will be performed. For the two secondary outcome variables that are measured in counts (i.e., ED attendance and the number of hospitalizations), GEE models with a log link function and a Poisson distribution will be performed. For the other secondary outcomes, which are continuous, GEE models with an identity link will be fitted. Significant time by group interactions in the GEE models will support our hypotheses on the effects of the e-health intervention using app support. Descriptive statistics will be used to summarize the level of satisfaction with the use of the app at T1 to T3 in the intervention group, and a GEE model will be used to assess changes in satisfaction over time. All of the tests will be two-sided and a p-value of <0.05 will be considered statistically significant.

This pilot study will examine the feasibility of the main RCT study by using the app,identify any recruitment, implementation of the intervention and logistic issues arising from the recruitment, intervention, and follow-ups. It can also provide the preliminary finding for sample size calculation for the main RCT later on.

ELIGIBILITY:
Inclusion Criteria:

* Chinese adults with a medical diagnosis of at-risk CHD disorders, including those with angina but no change in ST elevation on ECG and an acceptable troponin level 4 and those discharged from an ED; or those have at least two CHD risk factors : i) current regular smoker, ii) over 50 years of age; iii) has a medical diagnosis of diabetes or hypertension; iv) has a family history of ischaemic heart disease or hyperlipaedmia ;v) has hyperlipidaemia or is regularly taking drugs for hyperlipidaemia; vi) is obese (BMI>25); vii) has had a Percutaneous Coronary Intervention performed; and viii) was diagnosed with stable angina and prescribed with TNG drugs
* Those able to perform a brisk walking exercise and who have passed the 3-minute walking test
* Those who possess a smart phone and are able to use it.

Exclusion Criteria:

* Those with physical, mental, visual, or cognitive impairments for which they are undergoing regular medical follow-ups and treatment
* Those with musculoskeletal disorders or other disabling diseases that may limit the practice of any walking exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change of Self-efficacy and self-management behaviour | Baseline, 3 months
  Self-efficacy and self-management behaviour can be reflected by a total sum of score of a subscale of Self-efficacy in illness management (six items) and communication with healthcare professionals (three items) of the Self-Management Behaviour Questionnaire

SECONDARY OUTCOMES:
Blood pressure | 3 months
  systolic and diastolic blood pressure will be collected by trained research assistant.
Change of cardiovascular endurance test | Baseline, 3 months
  Three-minute step test aims to test the client's cardiovascular functional endurance after exercise across the age span and gender. A participant step on and off of a 12-inch high bench/ or stair for 3 minutes. Their pulse is then taken while the participant remains standing. Compare the heart rate with the table according to the age and gender to determine the fitness within a range of 7 scores from excellent to good, above average, average, below average, poor and very poor.
Change of total physical exercise | Baseline, 3 months
  This outcome will be measured using the Godin-Shepherd Leisure Time Physical Activity Questionnaire. This scale measures how often per week and how long per session the respondent has performed strenuous, moderate and mild exercise outside of their work duties.
Change of perceived stress scale (PSS-10) | Baseline, 3 months
  On this scale, 10 self-reported items are used to measure the degree to which situation in a person's life are considered stressful, as well as the current levels of stress experienced in the last month. The summative scores range from 0 to 40, with higher scores indicating higher stress levels. These scores have been used previously to assess the experienced level of stress as an outcome measure and have good psychometric properties in cardiac patients.
Change of Health literacy | Baseline, 3 months
  This outcome will be measured using 24-item Chinese Health Literacy Scale for Chronic Care (CHLCC). This scale has 4 sub scales: remembering, understanding, applying and analyzing. The total scores ranged from 0 to 48, and a higher total score indicates a higher level of health literacy. The CHLCC has good internal reliability ( Cronbach's α=0.91) and good test-retest reliability (intraclass correlation coefficient=0.77; p<0.01).
Change of Quality of Life:ED-5D | Baseline, 3 months
  The ED-5D is a generic instrument used to measure the quality of life in patients with cardiovascular disease in Chinese and other populations. These scale is divided into 5 parts: mobility, self-care, usual activities, pain/discomfort and anxiety/ depression. Participants are asked to respond to the items using the following options: no problem, moderate problems, and extreme problems. The 5 items will also be ranked on a visual analogue scale (VAS) with a range with points from 0 (worst possible health) to 100 (best possible health) to assess the patient's health. The ED-5D was found to be satisfactorily valid and reliable in many populations, including CHD patients.
Chest pain frequency | 3 months
  the frequency of chest pain attack will be record.
Satisfactory level of the programme | 3 months
  the satisfactory level will be asked with the scale 0-10
Hospitalization frequency | 3 months
  frequency of hospitalization will be asked.

OTHER OUTCOMES:
Change in body weight | baseline 3 months
  body weight will be measured at baseline and 3 months
Change in LDL cholesterol | baseline, 3 months
  Blood samples for measuring LDL cholesterol will be taken by using a finger stick using auto-analysed and the participants are asked to have 8 hours fasting.
Change in HDL cholesterol | baseline, 3 months
  Blood samples for measuring HDL cholesterol will be taken by using a finger stick using auto-analysed and the participants are asked to have 8 hours fasting.

CONTACTS AND LOCATIONS:
Overall Officials: Shuk Yee Ko, Principal Investigator — Tuen Mun Hospital; Lip Yip Lee, Principal Investigator — Tin Shui Wai Hospital
Locations (2):
- Hong Kong (2):
  - Tin Shui Wai Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong

REFERENCES:
- [Background] Lo SM, Choi KT, Wong EM, Lee LL, Yeung RS, Chan JT, Chair SY. Effectiveness of Emergency Medicine Wards in reducing length of stay and overcrowding in emergency departments. Int Emerg Nurs. 2014 Apr;22(2):116-20. doi: 10.1016/j.ienj.2013.08.003. Epub 2013 Aug 31. PMID 24080095
- [Background] Quan, X. [全晓丽 ]. (2017). The role of pain sensitivity, pain catastrophizing level and personality traits in influencing the pre-hospital delay of acute myocardial infarction patients. (Thesis). University of Hong Kong, Pokfulam, Hong Kong SAR.
- [Background] Lichtman JH, Froelicher ES, Blumenthal JA, Carney RM, Doering LV, Frasure-Smith N, Freedland KE, Jaffe AS, Leifheit-Limson EC, Sheps DS, Vaccarino V, Wulsin L; American Heart Association Statistics Committee of the Council on Epidemiology and Prevention and the Council on Cardiovascular and Stroke Nursing. Depression as a risk factor for poor prognosis among patients with acute coronary syndrome: systematic review and recommendations: a scientific statement from the American Heart Association. Circulation. 2014 Mar 25;129(12):1350-69. doi: 10.1161/CIR.0000000000000019. Epub 2014 Feb 24. PMID 24566200
- [Background] Tasić I, Lazarević G, Stojanović M, Kostić S, Rihter M, Djordjević D, et al. Health-related quality of life in patients with coronary artery disease after coronary revascularization. Central European Journal of Medicine. 2013;8(5):618-26.
- [Background] Artinian NT, Fletcher GF, Mozaffarian D, Kris-Etherton P, Van Horn L, Lichtenstein AH, Kumanyika S, Kraus WE, Fleg JL, Redeker NS, Meininger JC, Banks J, Stuart-Shor EM, Fletcher BJ, Miller TD, Hughes S, Braun LT, Kopin LA, Berra K, Hayman LL, Ewing LJ, Ades PA, Durstine JL, Houston-Miller N, Burke LE; American Heart Association Prevention Committee of the Council on Cardiovascular Nursing. Interventions to promote physical activity and dietary lifestyle changes for cardiovascular risk factor reduction in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 27;122(4):406-41. doi: 10.1161/CIR.0b013e3181e8edf1. Epub 2010 Jul 12. No abstract available. PMID 20625115
- [Background] Antypas K, Wangberg SC. An Internet- and mobile-based tailored intervention to enhance maintenance of physical activity after cardiac rehabilitation: short-term results of a randomized controlled trial. J Med Internet Res. 2014 Mar 11;16(3):e77. doi: 10.2196/jmir.3132. PMID 24618349
- [Background] Chow CK, Redfern J, Hillis GS, Thakkar J, Santo K, Hackett ML, Jan S, Graves N, de Keizer L, Barry T, Bompoint S, Stepien S, Whittaker R, Rodgers A, Thiagalingam A. Effect of Lifestyle-Focused Text Messaging on Risk Factor Modification in Patients With Coronary Heart Disease: A Randomized Clinical Trial. JAMA. 2015 Sep 22-29;314(12):1255-63. doi: 10.1001/jama.2015.10945. PMID 26393848
- [Background] Dang S, Karanam C, Gomez-Orozco C, Gomez-Marin O. Mobile Phone Intervention for Heart Failure in a Minority Urban County Hospital Population: Usability and Patient Perspectives. Telemed J E Health. 2017 Jul;23(7):544-554. doi: 10.1089/tmj.2016.0224. Epub 2017 Jan 4. PMID 28051761
- [Background] Dale LP, Whittaker R, Jiang Y, Stewart R, Rolleston A, Maddison R. Improving coronary heart disease self-management using mobile technologies (Text4Heart): a randomised controlled trial protocol. Trials. 2014 Mar 4;15:71. doi: 10.1186/1745-6215-15-71. PMID 24588893
- [Background] Khonsari S, Subramanian P, Chinna K, Latif LA, Ling LW, Gholami O. Effect of a reminder system using an automated short message service on medication adherence following acute coronary syndrome. Eur J Cardiovasc Nurs. 2015 Apr;14(2):170-9. doi: 10.1177/1474515114521910. Epub 2014 Feb 2. PMID 24491349
- [Background] Maddison R, Pfaeffli L, Whittaker R, Stewart R, Kerr A, Jiang Y, Kira G, Leung W, Dalleck L, Carter K, Rawstorn J. A mobile phone intervention increases physical activity in people with cardiovascular disease: Results from the HEART randomized controlled trial. Eur J Prev Cardiol. 2015 Jun;22(6):701-9. doi: 10.1177/2047487314535076. Epub 2014 May 9. PMID 24817694
- [Background] Piette JD, Striplin D, Marinec N, Chen J, Aikens JE. A randomized trial of mobile health support for heart failure patients and their informal caregivers: impacts on caregiver-reported outcomes. Med Care. 2015 Aug;53(8):692-9. doi: 10.1097/MLR.0000000000000378. PMID 26125415
- [Background] Pfaeffli Dale L, Whittaker R, Jiang Y, Stewart R, Rolleston A, Maddison R. Text Message and Internet Support for Coronary Heart Disease Self-Management: Results From the Text4Heart Randomized Controlled Trial. J Med Internet Res. 2015 Oct 21;17(10):e237. doi: 10.2196/jmir.4944. PMID 26490012
- [Background] Park LG, Howie-Esquivel J, Chung ML, Dracup K. A text messaging intervention to promote medication adherence for patients with coronary heart disease: a randomized controlled trial. Patient Educ Couns. 2014 Feb;94(2):261-8. doi: 10.1016/j.pec.2013.10.027. Epub 2013 Nov 18. PMID 24321403
- [Background] Wong EM, Chair SY, Leung DY, Sit JW, Leung KP. Home-based interactive e-health educational intervention for middle-aged adults to improve total exercise, adherence rate, exercise efficacy, and outcome: a randomised controlled trial. Hong Kong Med J. 2018 Feb;24 Suppl 2(1):34-38. No abstract available. PMID 29938656
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. PLoS Med. 2010 Mar 24;7(3):e1000251. doi: 10.1371/journal.pmed.1000251. PMID 20352064
- [Background] Kendall E, Catalano T, Kuipers P, Posner N, Buys N, Charker J. Recovery following stroke: the role of self-management education. Soc Sci Med. 2007 Feb;64(3):735-46. doi: 10.1016/j.socscimed.2006.09.012. Epub 2006 Oct 31. PMID 17079060
- [Background] Janz N, Champion V, Strecher V. The health belief model. In Glans K, RimerB, Lewis F, editors. Health behavior and health education -theory, research, and practice. 3rd ed. Jossey-Bass : John Wiley & Sons Inc.; 2002.
- [Background] Lin CH, Chiang SL, Tzeng WC, Chiang LC. Systematic review of impact of lifestyle-modification programs on metabolic risks and patient-reported outcomes in adults with metabolic syndrome. Worldviews Evid Based Nurs. 2014 Dec;11(6):361-8. doi: 10.1111/wvn.12069. PMID 25488565
- [Background] Siow E, Leung DYP, Wong EML, Lam WH, Lo SM. Do Depressive Symptoms Moderate the Effects of Exercise Self-efficacy on Physical Activity Among Patients With Coronary Heart Disease? J Cardiovasc Nurs. 2018 Jul/Aug;33(4):E26-E34. doi: 10.1097/JCN.0000000000000491. PMID 29851659
- [Background] Wong EM, Lo SM, Ng YC, Lee LL, Yuen TM, Chan JT, Chair SY. Cost-effectiveness of 'Program We Care' for patients with chronic obstructive pulmonary disease: A case-control study. Int Emerg Nurs. 2016 Jul;27:37-41. doi: 10.1016/j.ienj.2015.11.001. Epub 2015 Dec 2. PMID 26654881
- See also: World Health Organization. Cardiovascular diseases (CVDs). 2017. — http://www.who.int/mediacentre/factsheets/fs317/en/
- See also: Department of Health, The Hong Kong Special Administrative Region. Number of Deaths by Leading Causes of Death, 2001 - 2017. Department of Health, The Hong Kong Special Administrative Region — https://www.chp.gov.hk/en/statistics/data/10/27/117.html